CLINICAL TRIAL: NCT02892448
Title: Cardiac MRI for Metal on Metal Orthopaedic Prostheses
Brief Title: Cardiac MRI for Metal on Metal Hip Resurfacing
Acronym: CardiacMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20150281
Record Dates: First submitted 2016-08-04; First posted 2016-09-08 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-07

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral Hip Resurfacing (Active Comparator): Patients who received either right or left total hip resurfacing procedure. This group of patients will undergo a cardiac magnetic resonance imaging (CMR).
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)
- Bilateral Hip Resurfacing (Active Comparator): Patients who received both right and left hip resurfacing procedure on the same day. This group of patients will undergo a cardiac magnetic resonance imaging (CMR).
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)
- Non-Metal on Metal Total Hip (Active Comparator): Patients who received either a unilateral (one hip) or bilateral (both hips) non-metal on metal total hip arthroplasty. This group of patients will undergo a cardiac magnetic resonance imaging (CMR).
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)

INTERVENTIONS:
Other: Cardiac magnetic resonance imaging (CMR) — Cardiac MRI is used to assess cardiac function in patients at risk of cardiotoxicity. In addition, Cardiac MRI enables imaging of inflammation, and fibrosis in the heart which may provide more specific information about the mechanism of injury in patients with high ion blood levels. Patients in all three groups (Unilateral hip resurfacing, bilateral hip resurfacing, and non-metal on metal total hip arthroplasty) will undergo a Cardiac MRI.

SUMMARY:
There may be a relationship between heart function and the metal ion levels in patients having undergone total hip replacement. The idea is to use results from a clinical cardiac MRI to assess heart function in a sample of 30 patients whom have undergone either metal-on-metal hip replacement (unilateral or bilateral) or a non-metal on metal total hip replacement to determine whether having undergone a metal on metal hip procedure may be impacting heart function. In addition to the clinically used parameters, the images will also be retrospectively assessed using special software to assess amount of fibrosis and early changes affecting cardiac muscle contraction which may be indicative of impaired heart function. With these values we will compare to known, and previously collected, hip replacement and function data to determine whether there is any differences in how the heart works in those having had a hip replacement relative to a normal population.

DETAILED DESCRIPTION:
There has been some recent concern regarding possible systemic health effects resulting from elevated blood cobalt concentrations in patients with cobalt containing hip implants (1). To date there are no blood cobalt criteria to help guide physicians when evaluating an individual hip implant patient's risk of developing systemic health effects because historically there was little or no concern about systemic cobalt toxicity in implant patients. Included within this is heart function, for which investigators see a need to use this novel software to analyze heart function relative to Hip status and Metal Ion levels.

Patients with metal on metal hip prosthesis are subject to local and systemic release of cobalt and chromium ions which may increase the potential for locally aggressive ion-induced local tissue reactions such as pseudotumours, a type of Adverse Reaction to Metal Debris (ARMD) (2). Although there have been reports of local toxicity as well as cases of cobaltism (as seen during outbreak in Quebec of so called 'cobalt beer drinkers' cardiomyopathy) leading to cardiac and ototoxicity, it is unclear if chronic exposure to these ions can lead to impaired cardiac function (cardiotoxicity) in a well-functioning prosthesis.

The majority of the blood cobalt concentrations reported for hip implant patients appear to range from approximately 0.2 to 10 µg/L, and based on our review of the available literature, should not pose an increased risk for the development of systemic health effects.

The concern for systemic health effects is for the small number of patients with cobalt-containing hip implants with markedly elevated blood cobalt concentrations.

Extensive evaluations of these 'cobalt beer drinkers' have found that poor nutrition and underlying disease states caused by severe alcoholism were likely significant contributing factors to heart disease in this particular population. However, there remains a significant concern that cardiac function could be affected in the long term. This is especially relevant as the majority of these implants are put in patients less than 50 years age.

Cardiac magnetic resonance imaging (CMR) is the gold standard method to assess cardiac function in patients at risk of cardiotoxicity. In addition to assessing cardiac function, CMR enables imaging of inflammation, and fibrosis (which may be secondary to the ion deposition) in the heart which may provide more specific information about the mechanism of injury in these patients.

The purpose of this study is to look at cardiac function in patients with a metal on metal hip prostheses.

Recruitment: 30 patients in total (10 unilateral and 10 bilateral hip resurfacing patients and 10 non-metal on metal total hip replacement patients) will be recruited which should provide indication of relationship both between either instances and heart function, as well as compared to one another. All patients will be undergoing clinical cardiac MRI. All patients will have extra images collected during their MRI and these images will be analyzed to determine any relationship between heart function and the possible metal ion levels from the hip implant. As part of the scan analysis they will be required to also have a 5 millilitres (mLs) vial of blood collected. Ultrasound values will be retrospectively collected, for analysis of soft tissue reaction, from a previous clinically ordered ultrasound of the affected joint.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing clinical Cardiac MRI
* Currently enrolled with either unilateral or bilateral metal-on-metal (MoM) Hip replacement device
* Willing to sign Informed Consent Form

Exclusion Criteria:

* Patient does not meet all 'inclusion' criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- Paul E Beaule, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim PR, Beaule PE, Dunbar M, Lee JK, Birkett N, Turner MC, Yenugadhati N, Armstrong V, Krewski D. Cobalt and chromium levels in blood and urine following hip resurfacing arthroplasty with the Conserve Plus implant. J Bone Joint Surg Am. 2011 May;93 Suppl 2:107-17. doi: 10.2106/JBJS.J.01721. PMID 21543699
- [Background] Moon JC, Messroghli DR, Kellman P, Piechnik SK, Robson MD, Ugander M, Gatehouse PD, Arai AE, Friedrich MG, Neubauer S, Schulz-Menger J, Schelbert EB; Society for Cardiovascular Magnetic Resonance Imaging; Cardiovascular Magnetic Resonance Working Group of the European Society of Cardiology. Myocardial T1 mapping and extracellular volume quantification: a Society for Cardiovascular Magnetic Resonance (SCMR) and CMR Working Group of the European Society of Cardiology consensus statement. J Cardiovasc Magn Reson. 2013 Oct 14;15(1):92. doi: 10.1186/1532-429X-15-92. PMID 24124732
- [Background] Messroghli DR, Greiser A, Frohlich M, Dietz R, Schulz-Menger J. Optimization and validation of a fully-integrated pulse sequence for modified look-locker inversion-recovery (MOLLI) T1 mapping of the heart. J Magn Reson Imaging. 2007 Oct;26(4):1081-6. doi: 10.1002/jmri.21119. PMID 17896383
- [Background] Diesbourg LD, Prato FS, Wisenberg G, Drost DJ, Marshall TP, Carroll SE, O'Neill B. Quantification of myocardial blood flow and extracellular volumes using a bolus injection of Gd-DTPA: kinetic modeling in canine ischemic disease. Magn Reson Med. 1992 Feb;23(2):239-53. doi: 10.1002/mrm.1910230205. PMID 1549039
- [Result] Juneau D, Grammatopoulos G, Alzahrani A, Thornhill R, Inacio JR, Dick A, Vogel KI, Dobransky J, Beaule PE, Dwivedi G. Is end-organ surveillance necessary in patients with well-functioning metal-on-metal hip resurfacings? A cardiac MRI survey. Bone Joint J. 2019 May;101-B(5):540-546. doi: 10.1302/0301-620X.101B5.BJJ-2018-1478.R1. PMID 31039002

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
Started | 12 | 12 | 11
Completed | 10 | 10 | 10
Not Completed | 2 | 2 | 1
Not completed — Screening failure | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Full Range); unit: years] | 59.4 [52.2 to 66.5] | 57.7 [48.5 to 70.1] | 58.4 [51.8 to 70.2] | 58.5 [48.5 to 70.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 7
  Male | 9 | 8 | 6 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Time since implantation [Mean (Full Range); unit: years] | 9.1 [5.9 to 11.1] | 7.5 [6.7 to 9.1] | 6.7 [5.0 to 10.6] | 7.8 [5.0 to 11.1]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 28.1 [25.1 to 31.1] | 29.0 [25.3 to 34.4] | 27.1 [22.5 to 32.5] | 28.1 [22.5 to 34.4]
Body Surface Area (BSA) [Mean (Full Range); unit: m^2] | 2.04 [1.93 to 2.23] | 2.08 [1.79 to 2.32] | 1.97 [1.69 to 2.45] | 2.03 [1.69 to 2.45]

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Ejection Fraction
Description: The volumetric fraction of fluid ejected from a chamber with each contraction.
Time Frame: Minimum 5 years post-operative
Measure: Mean (Full Range); unit: Percent
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
Number analyzed (Participants) | 10 | 10 | 10
Percent
  Left ventricular ejection fraction | 64 [60 to 69] | 66 [63 to 72] | 65 [59 to 70]
  Right ventricular ejecton fraction | 62 [60 to 64] | 63 [58 to 70] | 62 [60 to 64]

2. Primary Outcome: Comprehensive Cardiac Function
Description: Volume measures including: left ventricular end-diastolic volume, left ventricular stroke volume, right ventricular end-diastolic volume, right ventricular end-systolic volume, right ventricular stroke volume
Time Frame: One time measure at CMR
Measure: Mean (Full Range); unit: mL/m^2
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
Number analyzed (Participants) | 10 | 10 | 10
mL/m^2
  Left ventricle end-diastolic volume (LVEDV) | 77 [68 to 80] | 73 [65 to 85] | 67 [61 to 70]
  Left ventricle end-systolic volume (LVESV) | 27 [20 to 39] | 26 [23 to 29] | 23 [19 to 29]
  Left ventricle stroke volume (LVSV) | 51 [42 to 56] | 46 [41 to 62] | 43 [41 to 46]
  Right ventricle end-diastolic volume (RVEDV) | 79 [76 to 87] | 82 [76 to 84] | 71 [64 to 77]
  Right ventricle end-systolic volume (RVESV) | 30 [22 to 35] | 30 [24 to 31] | 28 [22 to 31]
  Right ventricle stroke volume (RVSV) | 53 [46 to 57] | 50 [41 to 56] | 43 [41 to 46]

3. Primary Outcome: T2* Mapping Time
Description: T2* is a specific sequence in the cardiac MRI and mapping can lead to important indicators of cardiac structure and function.
Time Frame: One time measure at CMR
Measure: Mean (Full Range); unit: ms
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
Number analyzed (Participants) | 10 | 10 | 10
ms
  Myocardium | 32 [32 to 34] | 33 [32 to 34] | 33 [30 to 37]
  Liver | 27 [23 to 29] | 24 [15 to 26] | 28 [27 to 30]

4. Primary Outcome: T1 Mapping Time
Description: T1 is a specific sequence in the cardiac MRI and mapping can lead to important indicators of cardiac structure and function.
Time Frame: One time measure at CMR
Measure: Mean (Full Range); unit: ms
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
Number analyzed (Participants) | 10 | 10 | 10
ms
  Native T1 left ventricle (LV) average | 1003 [988 to 1014] | 988 [980 to 997] | 993 [987 to 1007]
  Post gadolinium T1 left ventricle (LV) average | 402 [384 to 432] | 409 [402 to 418] | 383 [371 to 397]

5. Secondary Outcome: Cobalt and Chromium Ion Levels
Description: To measure the level of cobalt and chromium ions in blood
Time Frame: Immediately Prior to cardiac MRI
Measure: Mean (Full Range); unit: ug/L
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
Number analyzed (Participants) | 10 | 10 | 10
ug/L
  Chromium blood levels | 1.41 [0.97 to 2.00] | 2.58 [1.60 to 2.90] | 0.11 [0.10 to 1.80]
  Cobat blood levels | 0.71 [0.50 to 1.07] | 1.47 [1.33 to 2.16] | 0.18 [0.16 to 0.19]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Unilateral Hip Resurfacing | Bilateral Hip Resurfacing | Non-Metal on Metal Total Hip
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT02892448/Prot_SAP_000.pdf